CLINICAL TRIAL: NCT07082803
Title: An Open-Label, Multicenter, Phase 1 Trial to Evaluate the Safety, Pharmacokinetics, and Anti-Tumor Activity of TLN-121 as a Single Agent and in Combination With Other Anti-Lymphoma Agents, in Patients With Relapsed or Refractory Non-Hodgkin Lymphomas
Brief Title: TLN-121 in Relapsed or Refractory Non-Hodgkin Lymphomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Treeline Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLN-121-2501
Record Dates: First submitted 2025-06-26; First posted 2025-07-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma; Lymphoma, Non Hodgkin
Keywords: Relapsed or Refractory Non-Hodgkin Lymphomas
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Agent (Experimental)
  Interventions: Drug: TLN-121
- Combination Treatment (Experimental)
  Interventions: Drug: TLN-254; Drug: TLN-121

INTERVENTIONS:
Drug: TLN-121 — Specified dose on specified days.
  Arms: Single Agent
Drug: TLN-254 — Specified dose on specified days.
  Arms: Combination Treatment
Drug: TLN-121 — Specified dose on specified days.
  Arms: Combination Treatment

SUMMARY:
The primary purpose of this study is to evaluate the safety, pharmacokinetics,, and preliminary anti-tumor activity of TLN-121 as a single agent and in combination with other anti-lymphoma therapies in patients with relapsed or refractory Non-Hodgkin Lymphomas

ELIGIBILITY:
Inclusion Criteria:

Disease Characteristics

1. Participant must have measurable disease at study entry
2. Participants must have one of the following histologically documented hematologic malignancies:

   1. Diffuse large B-cell lymphoma (DLBCL), not otherwise specified (DLBCL, NOS), Follicular lymphoma (FL) grade 3b, or transformed lymphoma from FL following at least 2 prior lines of therapy.
   2. FL grade 1-3a that requires treatment following at least 2 prior lines of therapy.
   3. The following Peripheral T-cell lymphoma (PTCL) subtypes that have relapsed after, or not responded to at least 1 prior systemic treatment regimen:

      * Nodal T-follicular helper (Tfh) cell lymphoma angioimmunoblastic; Follicular helper T-cell lymphoma, angioimmunoblastic type (AITL).
      * Nodal Tfh cell lymphoma, follicular type; Follicular helper T-cell lymphoma, follicular type.
      * Nodal Tfh cell lymphoma, NOS; Follicular helper T-cell lymphoma, NOS.
3. High-Grade B-Cell Lymphoma that has relapsed after, or not responded to at least 2 prior systemic treatment regimens.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

1. Participants must not have current central nervous system (CNS) involvement. Participants with past history of CNS involvement of lymphoma must have had CNS disease fully treated with no evidence of recurrence within 12 months.
2. Participant must not have a history of autologous stem cell transplantation within 60 days or allogeneic stem cell transplantation within 90 days prior to the start of the study.
3. Participant must not have a history of CAR T-cell or other T-cell targeting treatment ≤ 4 weeks prior to the start of the study.
4. Participant must not have major surgery or severe trauma within 4 weeks prior to the start of the study.
5. Participants must not have any condition, including significant acute or chronic medical illness, active or uncontrolled infection, or the presence of laboratory abnormalities, that places participants at unacceptable risk if participating in this study.
6. Pregnant or lactating.
7. Conditions that could affect drug absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing adverse events (AEs) that meet protocol-defined dose-limiting toxicity (DLT) criteria following administration of TLN-121 alone or in combination with TLN-254. | Up to 2 years
Incidence and Severity of Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related Adverse Events (TRAEs) | Up to 2 years
Clinically significant ECG QT Interval from baseline in safety laboratory test results, assessed as per NCI CTCAE v5.0 | Up to 2 years
Clinically significant laboratory abnormalities from baseline in safety laboratory test results, assessed as per NCI CTCAE v5.0 | Up to 2 years

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of TLN-121 | Up to 2 years
Time to Maximum Plasma Concentration (Tmax) of TLN-121 | Up to 2 years
Minimum Observed Plasma Concentration (Cmin) of TLN-121 | Up to 2 years
Area Under the Plasma Concentration-Time Curve (AUC) of TLN-121 | Up to 2 years
Anti-tumor activity of TLN-121 and TLN-121 in combination with TLN-254 by evaluating the objective response rate (ORR) according to the Lugano response criteria for Non-Hodgkin Lymphoma | Up to 2 years
Anti-tumor activity of TLN-121 and TLN-121 in combination with TLN-254 by evaluating the complete response rate (CR) according to the Lugano response criteria for Non-Hodgkin Lymphoma | Up to 2 years.
Anti-tumor activity of TLN-121 and TLN-121 in combination with TLN-254 by evaluating the duration of response (DOR) as assessed by the time from the date of first objective response to the date of disease progression | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (11):
- United States (5):
  - Stanford Medicine Cancer Center, Palo Alto, California
  - The START Center for Cancer Care - Midwest, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (5):
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Cabrini Health, Malvern, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Perth, Western Australia
- BC Cancer - Vancouver, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No